CLINICAL TRIAL: NCT00862576
Title: A Study of the Association of Sleep Dysfunction and Burning Mouth Syndrome
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Nita Chainani-Wu, Health Sciences Assistant Clinical Professor, University of California, San Francisco
Other Study IDs: H1113-29221
Record Dates: First submitted 2009-03-16; First posted 2009-03-17 (Estimated); Last update posted 2009-03-17 (Estimated); Status verified 2009-03

CONDITIONS: Burning Mouth Syndrome
Keywords: Burning Mouth Syndrome; Sleep; Neuropathic pain; Glossodynia; Chronic pain; Orofacial pain
MeSH Terms: conditions — Burning Mouth Syndrome; Neuralgia; Glossalgia; Chronic Pain; Facial Pain

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Burning Mouth Syndrome Group
- 2: Control Group

SUMMARY:
This is a case control study of the association between burning mouth syndrome and sleep dysfunction. Cases will comprise of patients diagnosed with burning mouth syndrome at the UCSF oral medicine clinic. Controls will include patients with leukoplakia, pigmented lesions, traumatic lesions, benign tumors, mucoceles, and pemphigoid matched on age (5 years) and gender to the cases. New patients as well as those presenting for follow-up visits will be eligible.

Each case and control subject will be administered the following 4 questionnaires by interview: (1) enrollment questionnaire (2) Sleep scale from the medical outcomes study (MOS), (3) current sleep status scale and (4) a numerical rating scale for measurement of oral symptoms.

Cases (BMS patients) will be followed in the clinic or by telephone contact once per month for the following 6 months and questionnaires 1 (question 6 only), 2, 3 and 4 will be administered by interview.

ELIGIBILITY:
Inclusion Criteria:

* Cases will comprise of patients diagnosed with burning mouth syndrome at the UCSF oral medicine clinic.
* Controls will include patients with leukoplakia, pigmented lesions, traumatic lesions, aphthous ulcers, reticular oral lichen planus, benign tumors, mucoceles, and pemphigoid matched on age (5 years) and gender to the cases.
* New patients as well as those presenting for follow-up visits will be eligible.

Exclusion Criteria:

* Age below 18 years
* Pregnancy
* Systemic corticosteroid therapy within the previous 2 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Seen at the Oral Medicine Clinic at the University of California, San Francisco
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2006-06; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Sleep quality and quantity

CONTACTS AND LOCATIONS:
Overall Officials: Nita Chainani-Wu, DMD, MS, PhD, Principal Investigator — University of California, San Francisco; Sol Jr. Silverman, MA, DDS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, California, United States